CLINICAL TRIAL: NCT01632553
Title: Longitudinal Measurement of Cortisol in Association With Mental Health and Experience of Domestic Violence and Abuse
Brief Title: Cortisol Evaluation in Abuse Survivors
Acronym: CEASE
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University College, London (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Survive South Gloucestershire and Bristol (Unknown)
Responsible Party: Principal Investigator, Gene Feder, Professor of Primary Health Care, Centre for Academic Primary Care, University of Bristol
Other Study IDs: 1678; NF110946 (Other Grant/Funding Number: Newton International Fellowships); SOCSRG2594 (Other: University of Bristol); insurance/CT1349 (Other: University of Bristol)
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Domestic Violence; Depression; Anxiety; Panic Disorder; Posttraumatic Stress Disorders
Keywords: Observation; Domestic Violence; Partner Abuse; Spousal Abuse; Battered Women; Abused Women; Cortisol; Mental Health; Depression; Anxiety; Posttraumatic Stress Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Panic Disorder; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: women who have experienced DVA
- Controls: women who have not experienced DVA

SUMMARY:
This study looks at the biological effect of domestic violence and abuse (DVA) on women's mental health. The mechanisms through which DVA causes mental disorders are very poorly understood. Similar to other demands, DVA activates the biological stress system, of which the chief component is the hypothalamic-pituitary-adrenal (HPA) axis, which produces chemical cortisol. Cortisol levels increase in response to short-term demand and help organisms deal with it by changing the processes of getting energy from food and also mental function. However constant activation of the HPA axis can cause damage and accelerate disease.

This study tests the hypothesis that compared to non-abused women all abuse victims have altered diurnal rhythm in cortisol secretion and that the pattern of this alteration is predicted by abuse characteristics, such as its type, severity, duration, and cessation. To examine the hypothesis the following research questions will be addressed: 1) whether cortisol levels are related to mental health state; 2) whether cortisol levels are related to type, severity, duration and cessation of DVA; 3) whether there is any difference in cortisol concentrations between those women exposed to both childhood abuse and DVA and those who have experienced only the latter; 4) whether cortisol levels vary between women, living in refuge and those not living in refuge?

To answer these research questions 214 women will be recruited in a domestic violence agency. Baseline and 3-monthly follow-up measures will be taken over 6 months after recruitment. Women will be asked to fill in a questionnaire to evaluate their demographics, health, experience of childhood abuse and DVA. Women's weight and height will be taken. In addition participants will be asked to take three saliva samples: 1st in the evening in bed, 2nd - next morning immediately upon awakening, and the 3rd - in thirty minutes after awakening. Saliva will be collected by chewing (for 2 minutes) the cotton pledget provided with plastic tube and returned by post or via collection by the researcher. Then the saliva samples will be tested for cortisol and cortisone.

Results of the study will increase our understanding of the biological mechanisms of DVA impact on a woman's health and tell researchers and practitioners about the possibility of using cortisol as an indicator to diagnose abuse-related health problems and assess effectiveness of medical care for abuse survivors.

DETAILED DESCRIPTION:
Domestic violence and abuse (DVA) is threatening behavior, violence or abuse (psychological, physical, sexual, financial or emotional) used by one person to control the other. Life time prevalence of DVA is 28% for women and 18% for men, although severity and consequences of abuse are less for men (1). Over and above damage to physical and reproductive health DVA has long-term detrimental effects on mental health for women consulting in primary care (2, 3). A meta-analysis of studies measuring the relationship between DVA and mental disorders reported increased risk for depression, anxiety, psychosomatic disorders, posttraumatic stress disorder (PTSD), alcohol abuse, and suicidal behavior (4). Kernic et al (5) have established that cessation of DVA among survivors is associated with decreased prevalence of depression; whereas Anderson and Sounders (6) have found that some women out of the abusive relationship may have greater psychological difficulties than those who are still in it. However the mechanisms through which DVA causes mental disease are very poorly understood. Similar to other stressors, DVA activates the biological stress system, of which the principal component is the hypothalamic-pituitary-adrenal (HPA) axis, which produces cortisol. Chronic activation of this system can result in dendritic retraction and hippocampal loss of function (7, 8). The results of existing cross-sectional studies testing the impact of DVA on women's HPA axis functioning are contradictory. Pico-Alfonso et al (9) have reported an increase in cortisol levels, whilst Seedat et al (10) have established reduction in cortisol levels in DVA subjects compared to controls. This disparity may relate to differential development of PTSD and/or depression within DVA-exposed samples (11). Currently, there is a hypothesis that DVA survivors may be characterized by alterations in the HPA axis (12) and that further longitudinal studies are needed to identify specific stress system disturbances in this group (1, 13). The aim of the study is to increase understanding of the role of hypothalamic-pituitary-adrenal (HPA) axis activity in DVA impact on women's mental health.

Study objectives:

* To evaluate the profiles of the awakening response of cortisol, the diurnal variation and the mean salivary cortisol concentration in women with experience of DVA and in non-abused controls
* To estimate whether cortisol secretion is associated with type, severity, duration and cessation of DVA
* To investigate whether cortisol acts as mediator between DVA and mental health state
* To examine whether there is any distinction in cortisol levels between those women exposed to both childhood abuse and DVA and those experienced only the latter
* To explore whether cortisol secretion differs between women, living in a domestic violence refuge/safe house and those still living in the community (after adjustment for confounding effects of abuse severity and continuing contact with abuser).

This 6-month study will consist of 3 measurements every 3 months. Each assessment will last approximately 30-45 minutes and will include:

1. Numerous standardized self-administered psychological questionnaires
2. Weight and height measurement
3. Self-completion of 3 saliva samples using Salivette tubes:

   1. evening sample - at bedtime
   2. awakening sample - in the morning immediately upon wakening
   3. post-awakening sample - 30 mins after awakening sample

Tubes with saliva will be returned by post or by researcher to an accredited laboratory for cortisol assay. The analysis also simultaneously measures cortisone a breakdown product of cortisol. This measurement is used to confirm the integrity of the sample.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 y.o.

Exclusion Criteria:

* unable to read English
* current use of steroid-based medications
* pregnancy
* presence of adrenal and/or pituitary gland disorder
* symptomatic psychotic illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women referred to two specialist domestic violence agencies for community outreach support or refuge accommodation by other agencies or self-referred. Non-abused friend and family controls will be recruited through index participants and in local communities through invitation letters displayed in public places in areas surrounding agencies sites.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Diurnal cortisol variation | Baseline, and at 3 and 6 months after baseline
  Difference between awakening and bedtime cortisol concentrations. Assay: Ultra performance liquid chromatography - tandem mass spectrometry (UPLC-MS/MS). Unit of measure - nmol/l.

SECONDARY OUTCOMES:
Cortisol awakening response (CAR) | Baseline, and at 3 and 6 months after baseline
  Difference between awakening and post awakening cortisol concentrations. Assay: UPLC - MS/MS. Unit of measure - nmol/l.
Mean salivary cortisol concentration | Baseline, and at 3 and 6 months after baseline
  Sum of awakening, post awakening, and bedtime cortisol concentrations. Assay: UPLC - MS/MS. Unit of measure - nmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Gene Feder, Professor, Principal Investigator — University of Bristol, Centre for Academic Primary Care; Stafford Lightman, Professor, Study Chair — University of Bristol, School of Clinical Sciences; Natalia Lokhmatkina, PhD, Study Director — University of Bristol, School of Clinical Sciences
Locations (2):
- United Kingdom (2):
  - Survive South Gloucestershire and Bristol, Kingswood, Bristol
  - Next Link, Bristol

REFERENCES:
- [Background] Feder G, Ramsay J, Dunne D, Rose M, Arsene C, Norman R, Kuntze S, Spencer A, Bacchus L, Hague G, Warburton A, Taket A. How far does screening women for domestic (partner) violence in different health-care settings meet criteria for a screening programme? Systematic reviews of nine UK National Screening Committee criteria. Health Technol Assess. 2009 Mar;13(16):iii-iv, xi-xiii, 1-113, 137-347. doi: 10.3310/hta13160. PMID 19272272
- [Background] Campbell JC. Health consequences of intimate partner violence. Lancet. 2002 Apr 13;359(9314):1331-6. doi: 10.1016/S0140-6736(02)08336-8. PMID 11965295
- [Background] Coid J, Petruckevitch A, Chung WS, Richardson J, Moorey S, Feder G. Abusive experiences and psychiatric morbidity in women primary care attenders. Br J Psychiatry. 2003 Oct;183:332-9; discussion 340-1. doi: 10.1192/bjp.183.4.332. PMID 14519611
- [Background] Golding JM. Intimate partner violence as a risk factor for mental disorders: A meta-analysis. Journal of Family Violence 14(2):99-132, 1999.
- [Background] Kernic MA, Holt VL, Stoner JA, Wolf ME, Rivara FP. Resolution of depression among victims of intimate partner violence: is cessation of violence enough? Violence Vict. 2003 Apr;18(2):115-29. doi: 10.1891/vivi.2003.18.2.115. PMID 12816399
- [Background] Anderson DK, Saunders DG. Leaving an abusive partner: an empirical review of predictors, the process of leaving, and psychological well-being. Trauma Violence Abuse. 2003 Apr;4(2):163-91. doi: 10.1177/1524838002250769. PMID 14697121
- [Background] Lightman SL. The neuroendocrinology of stress: a never ending story. J Neuroendocrinol. 2008 Jun;20(6):880-4. doi: 10.1111/j.1365-2826.2008.01711.x. PMID 18601712
- [Background] Mirescu C, Gould E. Stress and adult neurogenesis. Hippocampus. 2006;16(3):233-8. doi: 10.1002/hipo.20155. PMID 16411244
- [Background] Pico-Alfonso MA, Garcia-Linares MI, Celda-Navarro N, Herbert J, Martinez M. Changes in cortisol and dehydroepiandrosterone in women victims of physical and psychological intimate partner violence. Biol Psychiatry. 2004 Aug 15;56(4):233-40. doi: 10.1016/j.biopsych.2004.06.001. PMID 15312810
- [Background] Seedat S, Stein MB, Kennedy CM, Hauger RL. Plasma cortisol and neuropeptide Y in female victims of intimate partner violence. Psychoneuroendocrinology. 2003 Aug;28(6):796-808. doi: 10.1016/s0306-4530(02)00086-0. PMID 12812865
- [Background] McFarlane AC, Barton CA, Yehuda R, Wittert G. Cortisol response to acute trauma and risk of posttraumatic stress disorder. Psychoneuroendocrinology. 2011 Jun;36(5):720-7. doi: 10.1016/j.psyneuen.2010.10.007. Epub 2010 Nov 19. PMID 21093988
- [Background] Heim C, Ehlert U, Hanker JP, Hellhammer DH. Abuse-related posttraumatic stress disorder and alterations of the hypothalamic-pituitary-adrenal axis in women with chronic pelvic pain. Psychosom Med. 1998 May-Jun;60(3):309-18. doi: 10.1097/00006842-199805000-00017. PMID 9625218
- [Background] Dutton MA, Green BL, Kaltman SI, Roesch DM, Zeffiro TA, Krause ED. Intimate partner violence, PTSD, and adverse health outcomes. J Interpers Violence. 2006 Jul;21(7):955-68. doi: 10.1177/0886260506289178. PMID 16731994
- [Background] Lokhmatkina NV, Feder G, Blake S, Morris R, Powers V, Lightman S. Longitudinal measurement of cortisol in association with mental health and experience of domestic violence and abuse: study protocol. BMC Psychiatry. 2013 Jul 13;13:188. doi: 10.1186/1471-244X-13-188. PMID 23849084
- See also: protocol paper in Open Access — http://www.biomedcentral.com/1471-244X/13/188